CLINICAL TRIAL: NCT01369511
Title: A Phase 2 Randomized Study to Investigate the Efficacy and Safety of LY2495655 Versus Placebo in Older Patients Undergoing Elective Total Hip Arthroplasty
Brief Title: A Study of LY2495655 in Older Participants Undergoing Elective Total Hip Replacement
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11671; I1Q-MC-JDDE (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-06-07; First posted 2011-06-09 (Estimated); Results first posted 2018-06-06 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Muscular Atrophy
Keywords: Disuse Atrophy; Muscle; Strength; Arthroplasty; Hip; Joint Replacement
MeSH Terms: conditions — Muscular Atrophy; Muscular Disorders, Atrophic | interventions — landogrozumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Administered subcutaneously every 4 weeks for 12 weeks (administered 4 times)
  Interventions: Drug: Placebo
- 35 mg LY2495655 (Experimental): LY2495655: 35 milligrams (mg) administered subcutaneously every 4 weeks for 12 weeks (administered 4 times)
  Interventions: Drug: LY2495655
- 105 mg LY2495655 (Experimental): LY2495655: 105 mg administered subcutaneously every 4 weeks for 12 weeks (administered 4 times)
  Interventions: Drug: LY2495655
- 315 mg LY2495655 (Experimental): LY2495655: 315 mg administered subcutaneously every 4 weeks for 12 weeks (administered 4 times)
  Interventions: Drug: LY2495655

INTERVENTIONS:
Drug: LY2495655 — Administered subcutaneously
  Arms: 105 mg LY2495655; 315 mg LY2495655; 35 mg LY2495655
Drug: Placebo — Administered subcutaneously
  Arms: Placebo

SUMMARY:
The primary objective of this study is to test the hypothesis that appendicular lean body mass (aLBM) will increase after 12 weeks of LY2495655 treatment versus placebo in older participants undergoing elective total hip arthroplasty (eTHA).

ELIGIBILITY:
Inclusion Criteria:

* Males with a female partner of childbearing potential should use contraception during the treatment period of the trial and up to 15 weeks after the last dose of investigational product.
* Females should be of non-child bearing potential.
* Elective total hip arthroplasty (eTHA) is scheduled.
* Have a body mass index of <40 kilograms per square meter (kg/m^2) and a weight <136.4 kilograms (kg).
* Can climb at least 6 stairs with or without holding the handrail (but without human assistance), according to the participant at screening.
* Can stand up from a chair and walk more than 10 meters without human assistance.
* Takes at least 12 seconds to perform the Timed Up and Go (TUG) test at screening.

Exclusion Criteria:

* Another inpatient surgical procedure is planned in the 6 months following randomization.
* Lower extremity amputation.
* Lower-limb fracture within 6 months prior to screening or any major lower-limb surgery within 3 months prior to randomization.
* Simultaneous bilateral eTHA.
* The planned surgical procedure will preclude weight bearing for at least 4 weeks postoperatively (for instance, the planned procedure will involve extensive bone grafting). "Partial weight-bearing" and "weight-bearing as tolerated" are acceptable, but "non weight-bearing," "touch weight-bearing," or "feather weight-bearing" are exclusive.
* Underlying muscle disease (for example, polymyositis or muscular dystrophy) or a history of muscle disease other than age-associated muscle waste or disuse atrophy.
* Recent neurologic injury (<6 months prior to randomization) such as stroke or spinal cord injury, or unstable neurologic disorders that are likely to confound physical performance tests during the course of the study (such as unstable Parkinson disease or hemiplegia).
* History of positive testing for human immunodeficiency virus (HIV).
* Current use or previous use of any drugs known to influence muscle mass or performance within 6 months prior to randomization (this includes anabolic steroids, replacement therapy for gonadal deficiency, anti-androgens, luteinizing hormone-releasing hormone [LHRH] agonist and antagonists, growth hormone, Insulin-Like Growth Factor 1 [IGF1], or creatinine supplements) or systemic corticosteroid use for at least 3 months (in the last year) prior to randomization at a daily dose greater than or equal to a 10 mg prednisone equivalent.
* Severe Vitamin D deficiency defined as 25-hydroxy-vitamin D levels <9.2 nanograms per milliliter (ng/mL) or <23 nanomoles per milliliter (nmol/mL) at screening.
* History of a malignant neoplasm in the 5 years prior to screening, with the exception of superficial basal cell carcinoma or squamous cell carcinoma of the skin that has been definitively treated. Participants with carcinoma in situ of the uterine cervix treated definitively for more than 1 year prior to screening may enter the study.
* History of any of the following conditions within 90 days of screening: unstable angina, myocardial infarction, coronary artery bypass graft surgery, or percutaneous coronary intervention (such as, angioplasty or stent placement).
* Any current supraventricular arrhythmia with an uncontrolled ventricular response (mean heart rate >100 beats per minute [bpm]) at rest despite medical or device therapy, any history of spontaneous or induced sustained ventricular tachycardia (heart rate >100 bpm for 30 seconds) despite medical or device therapy, or any history of resuscitated cardiac arrest or the presence of an automatic internal cardioverter-defibrillator.
* Any history of congestive heart failure within 6 months of screening.
* Systolic blood pressure >160 or <90 millimeters of mercury (mmHg) or diastolic blood pressure >100 or <50 mmHg at screening, or malignant hypertension.
* An abnormality in the locally read 12-lead electrocardiogram (ECG) that in the opinion of the investigator increases the risk of participating in the study.
* Have either or both of the following: aspartate aminotransferase (AST), alanine aminotransferase (ALT) >2 times the upper limit of normal (ULN), or alkaline phosphatase >1.5 times ULN, or total bilirubin >1.5 times ULN.
* Known history or presence of severe acute or chronic liver disease.
* History of significant renal insufficiency, defined as receiving renal dialysis or having an estimated creatinine clearance <30 milliliters per minute (mL/minute) at screening.
* Current evidence or recent history of significant psychiatric disease such as dementia/Alzheimer's disease, schizophrenia, or bipolar disorder.
* Are currently enrolled in, or discontinued within the last 30 days (or 5 half-lives whichever is longer) from a clinical trial involving an investigational drug or off-label use of a drug, or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
* Regularly uses known drugs of abuse and/or shows positive findings on urinary drug screening (physician prescribed narcotics are allowed).
* Have a positive fecal occult blood (FOB) test at screening or cannot provide a stool sample for FOB testing prior to randomization.
* Have uncontrolled diabetes mellitus.
* Have had ocular trauma, ophthalmologic surgery, or eye laser treatment within 6 months prior to randomization.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2011-07; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY(1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST, Study Director — Eli Lilly and Company
Locations (45):
- United States (16):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tucson, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Laguna Hills, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lakewood, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Lauderdale, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pinellas Park, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gainesville, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boston, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Great Falls, Montana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wilmington, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Altoona, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., State College, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
- Austria (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vienna
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wiener Neustadt
- Belgium (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Genk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Merksem
- Canada (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newmarket, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Waterloo, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montreal, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Québec
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ballerup Municipality, Denmark
- Estonia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tallinn
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tartu
- Finland (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kuopio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oulu
- France (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cahors
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montauban
- Japan (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hokkaido
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wakayama
- Spain (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alzira
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Granada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
- Sweden (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stockholm
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Umeå
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Uppsala

REFERENCES:
- [Derived] Woodhouse L, Gandhi R, Warden SJ, Poiraudeau S, Myers SL, Benson CT, Hu L, Ahmad QI, Linnemeier P, Gomez EV, Benichou O; STUDY INVESTIGATORS. A Phase 2 Randomized Study Investigating the Efficacy and Safety of Myostatin Antibody LY2495655 versus Placebo in Patients Undergoing Elective Total Hip Arthroplasty. J Frailty Aging. 2016;5(1):62-70. doi: 10.14283/jfa.2016.81. PMID 26980371

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | 35 mg LY2495655 | 105 mg LY2495655 | 315 mg LY2495655
Started | 98 | 104 | 98 | 100
Received at Least 1 Dose of Study Drug | 98 | 103 (One participant was a screen failure and inadvertently randomized but did not receive study drug.) | 98 | 100
Completed | 85 | 91 | 87 | 89
Not Completed | 13 | 13 | 11 | 11
Not completed — Adverse Event | 1 | 1 | 5 | 0
Not completed — Entry criteria not met | 2 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1 | 2
Not completed — Protocol Violation | 0 | 1 | 0 | 2
Not completed — Physician Decision | 3 | 4 | 0 | 0
Not completed — Sponsor decision | 2 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 5 | 6 | 4 | 6

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- 35 mg LY2495655: LY2495655: 35 mg administered subcutaneously every 4 weeks for 12 weeks (administered 4 times)
- 105 mg LY2495666: LY2495655: 105 mg administered subcutaneously every 4 weeks for 12 weeks (administered 4 times)
- Total: Total of all reporting groups
Arm/Group | Placebo | 35 mg LY2495655 | 105 mg LY2495666 | 315 mg LY2495655 | Total
Number analyzed (Participants) | 98 | 104 | 98 | 100 | 400
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.38 (8.90) | 68.66 (8.09) | 67.85 (8.14) | 68.71 (7.95) | 68.65 (8.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 70 | 51 | 54 | 234
  Male | 39 | 34 | 47 | 46 | 166
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 0 | 2
  Not Hispanic or Latino | 52 | 51 | 56 | 55 | 214
  Unknown or Not Reported | 45 | 52 | 42 | 45 | 184
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 12 | 14 | 9 | 11 | 46
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 2 | 1 | 5
  White | 85 | 89 | 87 | 88 | 349
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  France | 0 | 3 | 0 | 1 | 4
  United States | 27 | 29 | 26 | 31 | 113
  Estonia | 11 | 5 | 13 | 12 | 41
  Canada | 16 | 20 | 19 | 19 | 74
  Finland | 7 | 4 | 7 | 4 | 22
  Belgium | 4 | 4 | 7 | 5 | 20
  Spain | 7 | 7 | 7 | 5 | 26
  Austria | 4 | 5 | 3 | 5 | 17
  Denmark | 11 | 11 | 6 | 6 | 34
  Japan | 11 | 14 | 9 | 11 | 45
  Sweden | 0 | 2 | 1 | 1 | 4
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per meter squared (kg/m^2)] — BMI was calculated by weight in kilograms divided by height in meters squared.
  kilograms per meter squared (kg/m^2) | 28.58 (4.82) | 28.78 (4.94) | 28.14 (4.31) | 28.51 (4.47) | 28.51 (4.63)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Appendicular Lean Body Mass (aLBM) at Week 12
Description: The percentage change in aLBM of 3 limbs (excluding the operated limb) was measured by dual energy x-ray absorptiometry (DEXA). Least squares (LS) means of the aLBM change from baseline to the 12 week endpoint was adjusted by baseline aLBM values as a covariate and treatment, visit, and the treatment-by-visit interaction were included as fixed effect via a mixed-effects model for repeated measured (MMRM) analysis.
Time Frame: Baseline, 12 Weeks
Population: Randomized participants with non-missing baseline and at least 1 post-baseline aLBM measure.
Measure: Least Squares Mean (Standard Error); unit: percentage change in aLBM (3 limbs)
Arm/Group | Placebo | 35 mg LY2495655 | 105 mg LY2495655 | 315 mg LY2495655
Number analyzed (Participants) | 70 | 68 | 76 | 69
percentage change in aLBM (3 limbs) | 0.297 (0.492) | 0.741 (0.500) | 1.018 (0.471) | 1.357 (0.494)
Statistical Analysis 1: Comparison: Placebo vs 35 mg LY2495655; at Week 12; Test type: Superiority or Other; p = 0.527, Mixed Models Analysis — p-values are from type 3 tests
Statistical Analysis 2: Comparison: Placebo vs 105 mg LY2495655; at Week 12; Test type: Superiority or Other; p = 0.291, Mixed Models Analysis — p-values are from type 3 tests
Statistical Analysis 3: Comparison: Placebo vs 315 mg LY2495655; at Week 12; Test type: Superiority or Other; p = 0.129, Mixed Models Analysis — p-values are from type 3 tests

2. Secondary Outcome: Change From Baseline in Appendicular Lean Body Mass (aLBM) at Weeks 4, 8, and 16
Description: The percentage change in aLBM of 3 limbs (excluding the operated limb) was measured by DEXA. LS means of the aLBM change from baseline to the 12 week endpoint was adjusted by baseline aLBM values as a covariate and treatment, visit, and the treatment-by-visit interaction were included as fixed effect via an MMRM analysis.
Time Frame: Baseline, 4 Weeks, 8 Weeks, and 16 Weeks
Population: Randomized participants with non-missing baseline and at least 1 post-baseline aLBM measure.
Measure: Least Squares Mean (Standard Error); unit: percentage change in aLBM (3 limbs)
Arm/Group | Placebo | 35 mg LY2495655 | 105 mg LY2495655 | 315 mg LY2495655
Number analyzed (Participants) | 74 | 69 | 80 | 72
percentage change in aLBM (3 limbs)
  Week 4 | NA (NA) — Data were not collected for this time point and not planned in the protocol because it was too close to the surgery date and associated swelling would confound results. | NA (NA) — Data were not collected for this time point and not planned in the protocol because it was too close to the surgery date and associated swelling would confound results. | NA (NA) — Data were not collected for this time point and not planned in the protocol because it was too close to the surgery date and associated swelling would confound results. | NA (NA) — Data were not collected for this time point and not planned in the protocol because it was too close to the surgery date and associated swelling would confound results.
  Week 8 | -0.900 (0.485) | -0.680 (0.498) | 0.340 (0.466) | 0.585 (0.488)
  Week 16: number analyzed (Participants) | 69 | 67 | 79 | 69
  Week 16 | -0.102 (0.494) | 0.606 (0.502) | 2.058 (0.467) | 1.784 (0.494)
Statistical Analysis 1: Comparison: Placebo vs 35 mg LY2495655; at Week 8; Test type: Superiority or Other; p = 0.751, Mixed Models Analysis — p-values are from type 3 tests
Statistical Analysis 2: Comparison: Placebo vs 105 mg LY2495655; at Week 8; Test type: Superiority or Other; p = 0.066, Mixed Models Analysis — p-values are from type 3 tests
Statistical Analysis 3: Comparison: Placebo vs 315 mg LY2495655; at Week 8; Test type: Superiority or Other; p = 0.031, Mixed Models Analysis — p-values are from type 3 tests
Statistical Analysis 4: Comparison: Placebo vs 35 mg LY2495655; at Week 16; Test type: Superiority or Other; p = 0.315, Mixed Models Analysis — p-values are from type 3 tests
Statistical Analysis 5: Comparison: Placebo vs 105 mg LY2495655; at Week 16; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis — p-values are from type 3 tests
Statistical Analysis 6: Comparison: Placebo vs 315 mg LY2495655; at Week 16; Test type: Superiority or Other; p = 0.007, Mixed Models Analysis — p-values are from type 3 tests

ADVERSE EVENTS:
Arm/Group | Placebo | 35 mg LY2495655 | 105 mg LY2495655 | 315 mg LY2495655
Serious Adverse Events (participants affected / at risk) | 14/98 | 8/104 | 16/98 | 3/100
Other Adverse Events (participants affected / at risk) | 72/98 | 76/104 | 66/98 | 68/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=98) | 35 mg LY2495655 (N=104) | 105 mg LY2495655 (N=98) | 315 mg LY2495655 (N=100)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device dislocation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Confusion postoperative (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint ankylosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1/47 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=98) | 35 mg LY2495655 (N=104) | 105 mg LY2495655 (N=98) | 315 mg LY2495655 (N=100)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 8 (8) | 7 (7) | 11 (11)
Constipation (Gastrointestinal disorders) | 8 (9) | 14 (15) | 7 (7) | 9 (9)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 8 (8) | 4 (4) | 5 (5)
Nausea (Gastrointestinal disorders) | 12 (12) | 20 (23) | 16 (18) | 21 (21)
Vomiting (Gastrointestinal disorders) | 9 (10) | 16 (20) | 9 (11) | 12 (12)
Fatigue (General disorders) | 7 (9) | 4 (4) | 4 (4) | 9 (9)
Injection site erythema (General disorders) | 0 (0) | 1 (1) | 2 (3) | 6 (11)
Injection site pain (General disorders) | 3 (3) | 6 (9) | 13 (30) | 12 (30)
Local swelling (General disorders) | 5 (5) | 6 (6) | 7 (7) | 3 (3)
Pyrexia (General disorders) | 11 (15) | 18 (22) | 13 (24) | 14 (14)
Influenza (Infections and infestations) | 6 (6) | 1 (1) | 2 (2) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 3 (4) | 2 (2) | 6 (7)
Urinary tract infection (Infections and infestations) | 3 (3) | 3 (4) | 3 (3) | 5 (6)
Anaemia postoperative (Injury, poisoning and procedural complications) | 2 (2) | 3 (4) | 2 (2) | 6 (6)
Oxygen saturation decreased (Investigations) | 7 (7) | 3 (3) | 3 (3) | 6 (6)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 1 (1) | 9 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (15) | 22 (30) | 11 (12) | 14 (23)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 9 (9) | 12 (14) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 9 (10) | 3 (4) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 11 (13) | 5 (6) | 4 (7)
Dizziness (Nervous system disorders) | 13 (16) | 9 (13) | 6 (7) | 9 (11)
Headache (Nervous system disorders) | 0 (0) | 6 (6) | 3 (4) | 2 (2)
Insomnia (Psychiatric disorders) | 3 (3) | 7 (7) | 7 (8) | 5 (5)
Urinary retention (Renal and urinary disorders) | 8 (8) | 5 (5) | 9 (9) | 8 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (8) | 3 (3) | 2 (2) | 3 (3)
Hypertension (Vascular disorders) | 6 (6) | 3 (3) | 3 (3) | 1 (1)
Hypotension (Vascular disorders) | 9 (11) | 9 (10) | 10 (10) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days